CLINICAL TRIAL: NCT05384119
Title: REVERT- Breast Cancer: Phase 1b/2 Study of the Addition of STAT3 Inhibitor TTI-101 to Reverse Resistance to Palbociclib or Ribociclib Plus Aromatase Inhibitor or Fulvestrant Therapy for Metastatic Hormone Receptor-Positive and HER2-Negative Breast Cancer
Brief Title: Phase 1b/2 Study of TTI-101 in Combination for Patients With Metastatic Hormone Receptor-Positive and HER2-Negative Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated prior to Phase 2 due to slow accrual.
Sponsor: Tvardi Therapeutics, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TVD-101-002B
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; HR+ HER2-, palbociclib-resistant breast cancer; TTI-101; STAT3 Inhibitor; Palbociclib; Aromatase inhibitor; ribociclib; fulvestrant
MeSH Terms: conditions — Breast Neoplasms | interventions — C188-9 compound; palbociclib; Aromatase Inhibitors; Fulvestrant; ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1b: Dose Escalation (Experimental): Participants will receive up to 3 dose levels of TTI-101 added to palbociclib and AI or fulvestrant to determine the RP2D.
  Interventions: Drug: TTI-101; Drug: Palbociclib; Drug: Aromatase inhibitor (AI); Drug: fulvestrant
- Phase 2: Dose Expansion (Experimental): Enrollment in Phase 2 may commence with approval from the safety review committee. Participants will be enrolled and treated at the RP2D of TTI-101 added to palbociclib or ribociclib and AI or fulvestrant.
  Interventions: Drug: TTI-101; Drug: Palbociclib; Drug: Aromatase inhibitor (AI); Drug: fulvestrant; Drug: ribociclib

INTERVENTIONS:
Drug: TTI-101 — Oral tablet
Drug: Palbociclib — Oral capsule
  Other Names: Ibrance ®
Drug: Aromatase inhibitor (AI) — Oral tablet
Drug: fulvestrant — Oral tablet
Drug: ribociclib — Oral tablet
  Arms: Phase 2: Dose Expansion

SUMMARY:
The primary objective of Phase 1b will be to evaluate the safety and tolerability of TTI-101 when added to palbociclib and AI or fulvestrant administered orally to participants with hormone receptor-positive (HR+) human epidermal receptor 2-negative (HER2)- palbociclib-resistant breast cancer, and to determine the recommended Phase 2 dose (RP2D) for TTI-101 when added to palbociclib and AI or fulvestrant.

The primary objective of Phase 2 will be to evaluate anti-tumor activity in participants who receive TTI-101 added to palbociclib or ribociclib and AI or fulvestrant.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following criteria to be eligible:

1. Age ≥18 years at the time of informed consent.
2. Metastatic or locally advanced breast cancer not amenable to curative treatment by surgery or radiotherapy.
3. For Phase 1b,currently receiving palbociclib and AI or fulvestrant; for Phase 2, currently receiving palbociclib or ribociclib and AI or fulvistrant therapy in the metastatic setting with evidence of progressive disease. In addition:

   * Must have remained on palbociclib or ribociclib and AI or fulvestrant therapy for ≥6 months for advanced breast cancer or metastatic disease prior to evidence of progression that in the opinion of the treating physician warrants continued therapy with palbociclib or ribociclib and AI or fulvestrant.
   * Dosage of palbociclib, ribociclib, AI and fulvestrant must remain unchanged from regimen prior to study enrollment specifically palbociclib at a dose of 125, 100, or 75 mg administered orally for 21 days every 28-day cycle or ribociclib at a dose of 200, 400, or 600 mg administered orally for 21 days every 28-day cycle.
4. All men and premenopausal women must be on medical gonadal suppression therapy with a gonadotropin analog (e.g, goserelin or leuprolide) and have estrogen levels in the postmenopausal range by institutional criteria at baseline.
5. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Has documented confirmation of histological or cytological HR-positive, HER2-negative breast cancer per local laboratory testing.
7. Up to 2 prior lines of systemic treatment (most recent line of therapy must be palbociclib and AI or fulvestrant for Phase 1b and palbociclib or ribociclib and AI or fulvestrant for Phase 2) in the locally advanced or metastatic setting is allowed; the participant must have shown evidence of progressive disease on palbociclib and AI or fulvestrant for Phase 1b and palbociclib or ribociclib and AI or fulvestrant for Phase 2 in the locally advanced or metastatic setting prior to enrollment.
8. Willing to provide a representative fresh tumor tissue specimen prior to enrollment. The fresh tumor specimen must be obtained after evidence of progression on palbociclib and AI or fulvestrant for Phase 1b and palbociclib or ribociclib and AI or fulvestrant for Phase 2.

   • Participants with bone only disease WITHOUT a soft tissue component, may opt out of the tumor biopsy.
9. The presence of measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 is preferred but not required. Lesions in a previously irradiated area that have not progressed are not considered measurable.

Exclusion Criteria:

Participants meeting any of the following exclusion criteria will not be eligible:

1. Has received more than 2 lines of prior systemic therapy for locally advanced/metastatic breast cancer.
2. Had prior exposure to any signal transducer and activator of transcription 3 (STAT3) inhibitor.
3. Had radiotherapy within 3 weeks prior to Cycle 1 Day 1 (cycle is 28 days). Participants must have recovered from radiotherapy toxicities prior to starting study treatment and recovered to Grade 1 or better from related side effects of such therapy (with the exception of alopecia).
4. Has HER2 overexpression by local laboratory testing (immunohistochemical [IHC] 3+ or in situ hybridization positive).
5. Has known loss of retinoblastoma tumor suppressor gene (Rb) (testing not mandatory).
6. Has had disease progression on more than two cyclin-dependent kinase (CDK)4/6 inhibitors. Adjuvant abemaciclib is allowed but must have progressed on palbociclib or ribociclib.
7. Concurrently using other anticancer therapy. Participants must continue palbociclib and AI or fulvestrant for Phase 1b and palbociclib or ribociclib and AI or fulvestrant for Phase 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Phase 1b: Number of Participants Who Experience a Dose Limiting Toxicity (DLT) | Day 1 to Day 28
Phase 1b: Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 18 months
  An AE is any untoward medical occurrence in a participant or clinical study participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Any clinically significant changes between baseline and postbaseline laboratory assessments, electrocardiograms (ECGs), vital signs and physical examinations will be recorded as AEs.
Phase 1b: Number of Participants Who Experience a Serious Adverse Event (SAE) | Up to approximately 18 months
Phase 2: Landmark Progression Free Sulrvival at 6 Months (PFS6) | Day 1 pre-dose and 6 months post-dose

SECONDARY OUTCOMES:
Phase 1b: PFS6 | Day 1 pre-dose and 6 months post-dose
Phase 1b and Phase 2: Clinical Benefit Rate (CBR) | Up to approximately 18 months
  Defined as complete response (CR) + partial response (PR) + stable disease (SD) for at least 6 months.
Phase 1b and Phase 2: Overall Response Rate (ORR) | Up to approximately 18 months
  Defined as complete response (CR) + partial response (PR) measured in all participants using RECIST Version 1.1.
Phase 1b and Phase 2: Overall Response Rate (ORR) | Up to approximately 18 months
  Defined as complete response (CR) + partial response (PR) measured using RECIST Version 1.1 in participants who have a follow-up on-study tumor assessment at least 42 days following Cycle 1 Day 1 (cycle is 28 days) and who receive at least 80% of scheduled dosing with TTI-101.
Phase 1b and Phase 2: Maximum Observed Plasma Concentration (Cmax) of TTI-101 | Cycle 2 Day 1 (cycle is 28 days)
Phase 1b and Phase 2: Time of Maximum Observed Plasma Concentration (Tmax) of TTI-101 | Cycle 2 Day 1 (cycle is 28 days)
Phase 1b and Phase 2: Area Under the Plasma Concentration-time Curve from Time 0 to Time t (AUC[0-t]) of TTI-101 | Cycle 2 Day 1 (cycle is 28 days)
Phase 1b and Phase 2: Pharmacodynamics of TTI-101 as Measured By Change from Baseline in Percentage of Phosphorylated Signal Transducer and Activator of Transcription 1 (pY-STAT1) Positive Cells in Tumor Biopsy Samples | Baseline to Cycle 3 Day 1 (cycle is 28 days)
Phase 1b and Phase 2: Pharmacodynamics of TTI-101 as Measured By Change from Baseline in Percentage of Phosphorylated Signal Transducer and Activator of Transcription 3 (pY-STAT3) Positive Cells in Tumor Biopsy Samples | Baseline to Cycle 3 Day 1 (cycle is 28 days)
Phase 1b and Phase 2: Pharmacodynamics of TTI-101 as Measured By Change from Baseline in Percentage of Phosphorylated Signal Transducer and Activator of Transcription 5 (pY-STAT5) Positive Cells in Tumor Biopsy Samples | Baseline to Cycle 3 Day 1 (cycle is 28 days)
Phase 1b and Phase 2: Duration of Response (DoR) to Treatment | Up to approximately 18 months
Phase 1b and Phase 2: Time to Tumor Progression (TTP) | Up to approximately 18 months
Phase 1b and Phase 2: Best Overall Response (BOR) | Up to approximately 18 months
Phase 2: Progression-free Survival (PFS) | Up to approximately 18 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Holy Cross Health Fort Lauderdale - Holy Cross Hospital, Fort Lauderdale, Florida
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - Vanderbilt - Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology - Dallas Fort Worth (DFW) - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Harold C. Simmons Comprehensive Cancer Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No